## Cover page with the Official Title of the study:

Behavioral Activation Therapy for Medical Students with Symptoms of Depression in Two Cities of Mexico

Date: May 1st of 2019

Informed Consent Form (ICF)





## **INFORMED CONSENT LETTER**

PROGRAM: BEHAVIORAL ACTIVATION THERAPY FOR MEDICAL STUDENTS WITH SYMPTOMS OF DEPRESSION IN TWO CITIES OF MEXICO.

| NAME OF THE PARTICIPANT: |
|-----------------------------------|
| DATE OF SIGNING INFORMED CONSENT: |
| NUMBER OF THE REGISTER: |

**Purpose:** The objective of the research is to validate the efficacy of a psychological treatment based on scientific evidence for the treatment of mild to moderate depression. As well as observing the modification of the alpha patterns in the brain activity.

**Procedure:** The study includes the application of various instruments oriented towards the detection of symptoms of depression such as:

- 1. EMOTIV EPOC + of 14 channels.
- 2. The Center for Epidemiologic Studies Depression (CES-D) scale.
- 3. The Depression, Anxiety and Stress Scale 21 Items (DASS-21).
- 4. Pittsburgh Sleep Quality Index
- 5. The Plutchik Suicide Risk Scale

You will receive a treatment based on the Behavioral Activation therapy, which includes the implementation of 8 modules distributed from 10 to 12 sessions, with a duration of one hour each.

Risks and Discomforts: No risk or discomfort has been detected in the participation in this research.

Confidentiality: The data of the participants will be treated with confidentiality, and destroyed once the study has concluded and after 5 years.

Benefits: Receive psychological treatment based on scientific evidence, without cost.

Participation: Your participation in this program is voluntary and can be withdrawn at any time you wish. If you wish to withdraw from the program, please notify the researcher in advance.

If you have any doubt, question or disagreement, you can clarify it with the person in charge of the project, Dr. Alejandro Domínguez Rodríguez, at his mail, alejandro.dominguez.rodriguez@uabc.edu.mx or MD. Jasshel Teresa Salinas-Saldivar at her email jasshel.salinas@uacj.mx.

| Name and signature of the participant. | Name and signature of who obtains the consent. |
|---|---|
| Witness 1. | Witness 2 |
| Name, address, relationship and signature | Name, address, relationship and signature |